CLINICAL TRIAL: NCT01877161
Title: Effects of Navigated Repetitive Transcranial Magnetic Stimulation According to Post-stroke Aphasia Types
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nam-Jong Paik, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: E-1206-158-003
Record Dates: First submitted 2013-03-11; First posted 2013-06-13 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-06

CONDITIONS: To Healthy Volunteer; Virtual Lesions for Aphasia

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Middle temporal gyrus (Experimental): Repetitive magnetic stimulation to middle temporal gyrus
  Interventions: Device: Repetitive magnetic stimulation to middle temporal gyrus
- Control group (Sham Comparator): Repetitive magnetic stimulation (Sham)
  Interventions: Device: Repetitive magnetic stimulation (Sham)
- Superior temporal gyrus (Experimental): Repetitive magnetic stimulation to superior temporal gyrus
  Interventions: Device: Repetitive magnetic stimulation to superior temporal gyrus

INTERVENTIONS:
Device: Repetitive magnetic stimulation to superior temporal gyrus — Repetitive magnetic stimulation to superior temporal gyrus
  Other Names: MagPro X100 magnetic stimulator
  Arms: Superior temporal gyrus
Device: Repetitive magnetic stimulation to middle temporal gyrus — Repetitive magnetic stimulation to middle temporal gyrus
  Other Names: MagPro X100 magnetic stimulator
  Arms: Middle temporal gyrus
Device: Repetitive magnetic stimulation (Sham) — Repetitive magnetic stimulation (Sham)
  Other Names: MagPro X100 magnetic stimulator
  Arms: Control group

SUMMARY:
Repetitive transcranial magnetic stimulation induced virtual lesions for aphasia.

DETAILED DESCRIPTION:
To evaluate the effect of navigated repetitive transcranial magnetic stimulation in subjects with aphasia after stroke.

ELIGIBILITY:
Inclusion Criteria:

* fluent in Korean
* older than 18 years old

Exclusion Criteria:

* younger than 18 years old
* psychotic or psychiatric problems
* pregnant
* contraindications to MRI/fMRI
* uncooperative
* metalic implants, pacemaker or cochlear implants
* cannot perform outcome measure-related task
* known seizure history

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nam-Jong Paik, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Bundang-gu, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period : 2012.12.05-2013.03.07 type of location: medical clinic through public announcement
Pre-assignment Details: 15 participants recruited: 15 screened, 0 excluded, 3 participants dropped out (3 participants withdrew because of their long-distance commute before group assignment)
Groups:
- rTMS Over MTG, STG, Sham: 3 sessions of Repetitive magnetic stimulation (rTMS) were applied to participants 3 sessions of rTMS were determined by a random sequence (eg. middle temporal gyrus (MTG)-superior temporal gyrus (STG)-Sham, Sham-MTG-STG, STG-MTG-Sham etc..0) The sequence of stimulation was counter-balanced across subjects.
  different sessions was performed after washout period (at least 3 days). The coil was placed perpendicularly to the scalp during sham rTMS sessions.
Period: First Session of Stimulation
Arm/Group | rTMS Over MTG, STG, Sham
Started | 12
Completed | 12
Not Completed | 0
Period: Washout (at Least 3 Days)
Arm/Group | rTMS Over MTG, STG, Sham
Started | 12
Completed | 12
Not Completed | 0
Period: Second Session of Stimulation
Arm/Group | rTMS Over MTG, STG, Sham
Started | 12
Completed | 12
Not Completed | 0
Period: Washout (at Least 3 Days)
Arm/Group | rTMS Over MTG, STG, Sham
Started | 12
Completed | 12
Not Completed | 0
Period: Third Session of Stimulation
Arm/Group | rTMS Over MTG, STG, Sham
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Same patients were stimulated over 2 different regions and with sham stimulation in a random order
Groups:
- rTMS Over MTG, STG, Sham: 3 sessions of Repetitive magnetic stimulation (rTMS) were applied to participants.
  3 sessions of rTMS were determined by a random sequence (eg. MTG-STG-Sham, Sham-MTG-STG, STG-MTG-Sham etc.) MTG: middle temporal gyrus STG: superior temporal gyrus
  The sequence of stimulation was counter-balanced across subjects. different sessions was performed after washout period (at least 3 days). The coil was placed perpendicularly to the scalp during sham rTMS sessions.
Arm/Group | rTMS Over MTG, STG, Sham
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 31.87 [24 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: The Change of Reaction Time Between Before and After Stimulation in Each Session (MTG, STG, Sham)
Description: Reaction time for lexical and repetition test were measured before and after the TMS stimulation at each sessions (at session 1, session 2, session 3 over MTG/STG/Sham; MTG: middle temporal gyrus, STG: superior temporal gyrus).
  Response times were measured via the response pad, and spoken responses were recorded via a SV-1 Voice Key apparatus.
  The "reaction time post TMS - reaction time pre TMS" were used for analysis.* Arm/Group Title Arm/Group Description Maximum length (999) Repetitive magnetic stimulation (rTMS) were applied over STG
Time Frame: change between before and after the TMS stimulation for each sessions (at session 1, session 2, session 3)
Measure: Mean (Standard Deviation); unit: msec
Groups:
- rTMS Over MTG: Repetitive magnetic stimulation (rTMS) were applied over MTG
- rTMS Over STG: Repetitive magnetic stimulation (rTMS) were applied over STG
- Sham rTMS: The coil was placed perpendicularly to the scalp during sham rTMS sessions.
Arm/Group | rTMS Over MTG | rTMS Over STG | Sham rTMS
Number analyzed (Participants) | 12 | 12 | 12
msec | 110.65 (102.97) | -14.25 (105.78) | 25.29 (109.74)

ADVERSE EVENTS:
Time Frame: during the stimulation and till the end of study participation
Arm/Group | Middle Temporal Gyrus | Control Group | Superior Temporal Gyrus
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No